CLINICAL TRIAL: NCT05632406
Title: Breathing & Blood Pressure
Status: Recruiting | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Other Study IDs: STUDY00003469
Record Dates: First submitted 2022-11-14; First posted 2022-11-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults without obesity: body mass index below 30 kg/m^2
- Adults with obesity: body mass index above 30 kg/m^2

SUMMARY:
The purpose of this study is to determine the effect of obesity on cardiovascular responses during various breathing maneuvers.

DETAILED DESCRIPTION:
Adults with higher body mass can have trouble breathing during exercise, which could be due to high respiratory muscle workloads. These breathing muscles can require a lot of energy, which takes away energy from other (e.g., leg) muscles. Participating in this study will help us understand how the heart and blood vessels respond during brief exercise and during various breathing maneuvers.

ELIGIBILITY:
Inclusion Criteria:

• Body mass index values of ≤40 kg/m^2

Exclusion Criteria:

* Not weight stable (<5% change in body mass over the past six months)
* Overt cardiovascular, neurological, renal, liver, and/or metabolic illness (e.g., diabetes mellitus)
* Current, or history of uncontrolled, Stage 2 hypertension (blood pressure >140 / 90 mmHg; anti-hypertensive medications are permitted)
* Diagnosed obstructive sleep apnea
* Previous bariatric surgery
* Diagnosis or signs (e.g., values below the lower limit of normal) of overt airway disease(s)
* Current or recent (regular use within the past 6 months) use of tobacco or nicotine products (e.g., cigarettes, vaping)
* Per the POWERbreathe® company:
* Patients who have undergone recent abdominal surgery and those with abdominal hernia.
* Asthma patients who have a very low symptom perception and suffer from frequent, severe exacerbations or with an abnormally low perception of dyspnoea.
* If a patient is suffering from a ruptured eardrum or any other condition of the ear.
* Patients with marked elevated left ventricular end-diastolic volume and pressure.
* Patients with worsening heart failure signs and symptoms after a respiratory/inspiratory muscle training (IMT) session
* If you are suffering from a cold, sinusitis, or respiratory tract infection, we advise that you do not use your POWERbreathe IMT device.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant (self-reported and urine pregnancy test conducted), lactating (self-reported), or post-menopausal (self-reported) females
* Prisoners

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals living in, or near, Tallahassee, FL, USA
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure during exercise | Up to one week
  Systolic and diastolic blood pressure measured in the laboratory at rest and during an incremental aerobic exercise test

SECONDARY OUTCOMES:
Blood pressure during respiratory muscle testing | Up to one week
  Systolic and diastolic blood pressure measured in the laboratory at rest and during a respiratory muscle exercise test (eucapnic voluntary hyperpnea)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Watso, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate data and/or material transfer agreement approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of the trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of appropriate data and/or material transfer agreement approvals with the study PI and their institution.

REFERENCES:
- See also: Related Info — http://caplaboratory.com